CLINICAL TRIAL: NCT00564681
Title: Study to Evaluate Safety, Efficacy of Botulinum Toxin Type A in Patients With Cervical Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-090
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- botulinum toxin Type A (Active Comparator): Intramuscular injections into the affected muscles. Maximum dose of 360 units. Subjects may receive up to three treatments.
  Interventions: Biological: botulinum toxin type A
- botulinum toxin Type A Formulation 2 (Active Comparator): Intramuscular injections into the affected muscles. Maximum dose of 360 units. Subjects may receive up to three treatments.
  Interventions: Biological: botulinum toxin type A Formulation 2
- Placebo (Normal Saline) / botulinum toxin Type A (Other): Intramuscular injections of the assigned study medication into the affected muscles (placebo for treatment cycle 1 and botulinum toxin Type A for subsequent treatments). Maximum dose of 360 units. Subjects may receive up to three treatments.
  Interventions: Biological: botulinum toxin type A; Drug: Normal Saline
- Placebo (Normal Saline) / botulinum toxin Type A Formulation 2 (Other): Intramuscular injections of the assigned study medication into the affected muscles (placebo for treatment cycle 1 and botulinum toxin Type A Formulation 2 for subsequent treatments). Maximum dose of 360 units. Subjects may receive up to three treatments.
  Interventions: Biological: botulinum toxin type A Formulation 2; Drug: Normal Saline

INTERVENTIONS:
Biological: botulinum toxin type A — Intramuscular injections into the affected muscles. Maximum dose of 360 units. Subjects may receive up to three treatments.
  Other Names: BOTOX®
  Arms: Placebo (Normal Saline) / botulinum toxin Type A; botulinum toxin Type A
Biological: botulinum toxin type A Formulation 2 — Intramuscular injections into the affected muscles. Maximum dose of 360 units. Subjects may receive up to three treatments.
  Arms: Placebo (Normal Saline) / botulinum toxin Type A Formulation 2; botulinum toxin Type A Formulation 2
Drug: Normal Saline — Intramuscular injections of placebo (normal saline) into the affected muscles for treatment cycle 1.
  Arms: Placebo (Normal Saline) / botulinum toxin Type A; Placebo (Normal Saline) / botulinum toxin Type A Formulation 2

SUMMARY:
Study is to investigate the use of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale in a cervical dystonia population treated with botulinum toxin type A, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical dystonia

Exclusion Criteria:

* Current or previous botulinum toxin treatment of any type for any condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (16):
- Winston-Salem, North Carolina, United States
- Halifax, Nova Scotia, Canada
- Prague, Czechia
- Berlin, Germany
- Budapest, Hungary
- Mumbai, India
- Manila, Philippines
- Warsaw, Poland
- Moscow, Russia
- Belgrade, Serbia
- Singapore, Singapore
- Spisska Nova, Slovakia
- Cape Town, South Africa
- Tainan, Taiwan
- Bangkok, Thailand
- Bristol, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline) / Botulinum Toxin Type A | Placebo (Normal Saline) / Botulinum Toxin Type A Formulation 2
Started | 117 | 61 | 43 | 21
Completed | 106 | 58 | 40 | 19
Not Completed | 11 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline) / Botulinum Toxin Type A | Placebo (Normal Saline) / Botulinum Toxin Type A Formulation 2 | Total
Number analyzed (Participants) | 117 | 61 | 43 | 21 | 242
Age, Customized [Number; unit: Participants]
  <45 years | 38 | 22 | 13 | 11 | 84
  Between 45 and 65 years | 71 | 28 | 24 | 8 | 131
  >65 years | 8 | 11 | 6 | 2 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 43 | 32 | 13 | 169
  Male | 36 | 18 | 11 | 8 | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Observed Total Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Score at Week 4 of Treatment Cycle 1
Description: Change from baseline in observed TWSTRS score at Week 4 of Treatment Cycle 1. The TWSTRS is an assessment scale used to measure the impact of cervical dystonia on patients. The score is comprised of 3 subscales: Severity, Disability, and Pain, each of which is scored independently. The total of these 3 comprises the TWSTRS total score which is scored from 0 (least symptoms) to 85 (worst symptoms). Higher scores indicate a greater degree of symptom severity. A negative change from baseline represents improvement and a positive change from baseline indicates worsening.
Time Frame: Baseline, Week 4
Population: Intent-To-Treat: All enrolled patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Botulinum Toxin Type A; Botulinum Toxin Type A Formulation 2: Intramuscular injections into the affected muscles. Maximum dose of 360 units.
- Placebo (Normal Saline): Intramuscular injections into the affected muscles. Includes all patients who received placebo in Cycle 1.
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline)
Number analyzed (Participants) | 117 | 61 | 64
Scores on a Scale
  Baseline | 40.4 (9.14) | 41.5 (9.40) | 39.6 (9.52)
  Change from Baseline at Week 4 | -10.3 (9.77) | -13.6 (10.20) | -5.6 (8.58)

2. Secondary Outcome: Physician's Global Assessment of Response to Treatment at Week 4 of Treatment Cycle 1
Description: Physician's global assessment of response to treatment at Week 4 of Treatment Cycle 1. Responses were measured on a 9-point scale of +4 to -4, with higher scores denoting improvement in cervical dystonia: +4 was 'Complete abolishment of signs and symptoms (100% improvement)', 0 represented 'No change', and -4 represented 'Very marked worsening (about 100% worse or greater)'.
Time Frame: Week 4
Population: Intent-to-Treat: All enrolled patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline)
Number analyzed (Participants) | 117 | 61 | 64
Scores on a Scale | 1.3 (1.13) | 1.6 (1.04) | 0.8 (1.00)

3. Secondary Outcome: Patient's Global Assessment of Response to Treatment at Week 4 of Treatment Cycle 1
Description: Patient's global assessment of response to treatment at Week 4 of Treatment Cycle 1. Responses were measured on a 9-point scale of +4 to -4, with higher scores denoting improvement in cervical dystonia: +4 was 'Complete abolishment of signs and symptoms (100% improvement)', 0 represented 'No change', and -4 represented 'Very marked worsening (about 100% worse or greater)'.
Time Frame: Week 4
Population: Intent-to-Treat: All enrolled patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline)
Number analyzed (Participants) | 117 | 61 | 64
Scores on a Scale | 1.3 (1.31) | 1.5 (1.07) | 0.6 (1.06)

4. Secondary Outcome: Change From Baseline in Pain as Evaluated With the TWSTRS Pain Subscale at Week 4 of Treatment Cycle 1
Description: Change from baseline in pain as evaluated with the TWSTRS pain subscale at Week 4 of Treatment Cycle 1. The TWSTRS pain subscale scores range from 0 to 20 (0=no pain and 20=worst pain), based on severity of neck pain (0=no pain and 10=worst pain), the duration of pain (0=none and 5=most), and the degree of disability (0=none and 5=most). A negative number change from Baseline represents a decrease in pain (improvement).
Time Frame: Baseline, Week 4
Population: Intent-to-Treat: All enrolled patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline)
Number analyzed (Participants) | 117 | 61 | 64
Scores on a Scale
  Baseline | 9.7 (4.04) | 10.0 (3.41) | 9.7 (4.13)
  Change from Baseline at Week 4 | -2.8 (3.72) | -4.1 (4.15) | -1.3 (3.59)

5. Secondary Outcome: Duration of Treatment Effect for Treatment Responders
Description: Duration of Treatment Effect for Treatment Responders is defined as the number of days from the date of first treatment to the first visit after Week 4 of Treatment Cycle 1, at which the Total TWSTRS score reaches at least 90% of the baseline score. A treatment responder is defined as a patient who has at least a 30% reduction in Total TWSTRS score at Week 4 after the first treatment. The TWSTRS score measures the impact of cervical dystonia on patients (0=least symptoms and 85= worst symptoms).
Time Frame: Up to 6 Months
Population: Intent-to-Treat: All enrolled patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline)
Number analyzed (Participants) | 117 | 61 | 64
Days | 111.0 [97.00 to 119.00] | 99.0 [96.00 to 113.00] | 99.0 [92.00 to 109.00]

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for serious adverse events (SAEs) and adverse events (AEs) and is the total number of patients that were randomized AND treated. SAEs and AEs are presented by randomized arm and not necessarily by treatment received.
Arm/Group | Botulinum Toxin Type A | Botulinum Toxin Type A Formulation 2 | Placebo (Normal Saline) / Botulinum Toxin Type A | Placebo (Normal Saline) / Botulinum Toxin Type A Formulation 2
Serious Adverse Events (participants affected / at risk) | 9/117 | 1/61 | 5/42 | 1/21
Other Adverse Events (participants affected / at risk) | 83/117 | 41/61 | 31/42 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=117) | Botulinum Toxin Type A Formulation 2 (N=61) | Placebo (Normal Saline) / Botulinum Toxin Type A (N=42) | Placebo (Normal Saline) / Botulinum Toxin Type A Formulation 2 (N=21)
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=117) | Botulinum Toxin Type A Formulation 2 (N=61) | Placebo (Normal Saline) / Botulinum Toxin Type A (N=42) | Placebo (Normal Saline) / Botulinum Toxin Type A Formulation 2 (N=21)
Neck Pain (Musculoskeletal and connective tissue disorders) | 20 | 10 | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19 | 2 | 4 | 5
Dysphagia (Gastrointestinal disorders) | 10 | 7 | 4 | 2
Injection site pain (General disorders) | 9 | 5 | 3 | 4
Hypertension (Vascular disorders) | 8 | 3 | 1 | 0
Headache (Nervous system disorders) | 7 | 6 | 4 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 2 | 3
Nausea (Gastrointestinal disorders) | 6 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 3
Influenza-like illness (General disorders) | 2 | 2 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 0
Influenza (Infections and infestations) | 1 | 2 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo